CLINICAL TRIAL: NCT06564246
Title: Clinical Study Evaluating The Role of Vonoprazan Versus Pantoprazole in Patients With Gastroesophageal Reflux Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Aya Hany Abdelaziz Fahmy, Master degree student at faculty of pharmacy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT(829)
Record Dates: First submitted 2024-08-18; First posted 2024-08-21 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: Vonoprazan; Pantoprazole; Gastroesophageal Reflux Disease (GERD); Gastrin serum level; E-Cadherin level
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Intervention Model Description: * Group 1 (control group): 22 patients who will receive Vonoprazan 20mg (Vonseca) and placebo of pantoloc daily for 8 weeks.
  * Group 2: 22 patients who will receive Pantoprazole 40 mg (Pantoloc) and placebo of vonseca daily for 8 weeks.
Who Masked: Participant
Masking Description: single blinded study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vonoprazan 20mg (Vonseca) (Active Comparator): • Group 1 (control group): 22 patients who will receive Vonoprazan 20mg (Vonseca) and placebo of pantoprazole (pantoloc) daily for 8 weeks
  Interventions: Drug: Vonoprazan 20 mg versus Pantoprazole 40 mg
- Pantoprazole 40 mg (Pantoloc) (Active Comparator): • Group 2: 22 patients who will receive Pantoprazole 40 mg (Pantoloc) and placebo of vonoprazan (vonseca) daily for 8 weeks.
  Interventions: Drug: Vonoprazan 20 mg versus Pantoprazole 40 mg

INTERVENTIONS:
Drug: Vonoprazan 20 mg versus Pantoprazole 40 mg — Patients divided into two arms First Arm administered vonoprazan Second arm administered pantoprazole
  Other Names: Vononoprazan (Vonesca) versus pantoprazole (pantoloc)

SUMMARY:
This study aims to investigate the possible efficacy of vonoprazan versus Pantoprazole in patients with gastroesophageal reflux disease.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) occurs when stomach acid repeatedly flows back into the esophagus with or without histological changes. However, the excessive reflux of gastric acid induces some complications, such as esophagitis, esophageal stenosis, cancer or Barrett's esophagus. GERD is classified into two categories: nonerosive reflux disease (NERD) and erosive esophagitis. NERD is characterized by the presence of the typical symptoms of GERD without visible erosive esophagitis on endoscopy. Erosive esophagitis is characterized by injury to the esophageal mucosa on endoscopy. The major symptoms of GERD include heartburn, acid regurgitation and decrease the patient's quality of life (QOL). Therefore, improvement in the QOL of these patients by supplying rapid relief of symptoms is the primary objective of treatment.

For decades, proton pump inhibitors (PPIs) have been the mainstay of treatment for erosive esophagitis. Long-term maintenance therapy with PPIs is also recommended to keep healing in patients with more severe erosive esophagitis, given that recurrence occurs in nearly 100% of such patients without therapy. Furthermore, PPIs are restricted in their time of dosing. PPIs are prodrugs that are converted to their active form in the acidic environment of the secretory canaliculus, which is also the sole location of active proton pumps in the parietal cell. Thus, PPIs only inhibit active proton pumps. Given their limited duration of action (half-life nearly 1-2 hours), PPI are taken 30 to 60 minutes before a meal so their presence in the secretory canaliculus coincides with the postprandial peak in active proton pumps.

An alternative therapy for patients who may not respond to PPIs and that does not have the requirement for dosing around meals might be of utility. Such a potential alternative therapy is a potassium competitive acid blocker (PCAB), a new class of antisecretory agent that supplies more potent inhibition of gastric acid than PPI.

PCAB exhibits a more rapid onset of action than PPIs and achieves a maximum acid inhibitory effect on the 1st day after treatment, while PPIs require 3-5 days. However, few studies have examined whether the rapid onset of vonoprazan contributes to the clinical effects on the typical GERD symptoms of heartburn and acid regurgitation.

The previously mentioned findings highlight the need for further studies to evaluate the role of vonoprazan in patients with gastroesophageal reflux disease.

Aim of the Work The aim of this study is to investigate the possible efficacy of vonoprazan versus Pantoprazole in patients with gastroesophageal reflux disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 17-60 years.
* Both genders.
* Patients with a score ≥ 8 on the Gastroesophageal Reflux Disease Questionnaire (Gerd Q) are defined as having GERD and will enroll in this study and it will be done at baseline and after 8 weeks.

Exclusion Criteria:

* Subjects with history of gastrointestinal disease, gastroduodenal surgery, inflammatory bowel disease and Barrett's esophagus.
* Subjects with an earlier or current history of Zollinger-Ellison syndrome, or other gastric acid hypersecretion disorders (gastric or duodenal ulcer).
* Subjects with history of total/subtotal gastrectomy and esophageal achalasia.
* Subjects with Corona virus disease (COVID19).
* Subjects with major cardiological, respiratory, endocrine metabolic disease and neuro-psychological disease.
* Pregnancy or lactation.
* Subjects with total bilirubin level ≥ 1.2 mg/dl and ALT level > 100 IU/l.
* Subjects with renal impairment (Crcl less than 30 ml/min).
* Patients receiving atazanavir sulphate, nelfinavir and rilpivirine hydrochloride due to potential drug interactions.

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
change in the measured biomarker | Before and after 2 months
  Measured biomarkers are serum gastrin hormone and E-Cadherin level

SECONDARY OUTCOMES:
Change in gastroesophageal reflux disease symptoms (The Structured Assessment of Gastrointestinal Symptoms Questionnaire). | Before and after 2 months
  Structured Assessment of Gastrointestinal Symptoms Scale (SAGIS) is a validated measure of the intensity and impact of 22 upper and lower gastrointestinal symptoms. Responses are given on a 5 point Likert scale from no problem, mild (can be ignored when you do not think about it), moderate (cannot be ignored, but does not influence daily activities), severe (influencing your concentration on daily activities) and very severe (markedly influences your daily activities
  &/or requires rest) problem. In addition the SAGIS asks about the presence of selected non gastrointestinal symptoms including headache, chronic fatigue, back pain, sleep disturbances, depression and anxiety. The patient also answers the following questions, "In your own words, what is your most important health concern or problem?" and "In your own words, what is your second most important health concern or problem?

CONTACTS AND LOCATIONS:
Overall Officials: Aya Hany Abdel Aziz, Principal Investigator — Master degree student at faculty of pharmacy - Tanta university
Locations (1):
- Theodore Billiharz Institute for Researchs, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim YS, Kim TH, Choi CS, Shon YW, Kim SW, Seo GS, Nah YH, Choi MG, Choi SC. Effect of itopride, a new prokinetic, in patients with mild GERD: a pilot study. World J Gastroenterol. 2005 Jul 21;11(27):4210-4. doi: 10.3748/wjg.v11.i27.4210. PMID 16015691
- [Background] Sakurai K, Suda H, Fujie S, Takeichi T, Okuda A, Murao T, Hasuda K, Hirano M, Ito K, Tsuruta K, Hattori M. Short-Term Symptomatic Relief in Gastroesophageal Reflux Disease: A Comparative Study of Esomeprazole and Vonoprazan. Dig Dis Sci. 2019 Mar;64(3):815-822. doi: 10.1007/s10620-018-5365-0. Epub 2018 Nov 10. PMID 30415407
- [Background] Altomare A, Guarino MP, Cocca S, Emerenziani S, Cicala M. Gastroesophageal reflux disease: Update on inflammation and symptom perception. World J Gastroenterol. 2013 Oct 21;19(39):6523-8. doi: 10.3748/wjg.v19.i39.6523. PMID 24151376
- [Background] Armstrong D. Endoscopic evaluation of gastro-esophageal reflux disease. Yale J Biol Med. 1999 Mar-Jun;72(2-3):93-100. PMID 10780570
- [Background] Hongo M, Kinoshita Y, Miwa H, Ashida K. The demographic characteristics and health-related quality of life in a large cohort of reflux esophagitis patients in Japan with reference to the effect of lansoprazole: the REQUEST study. J Gastroenterol. 2008;43(12):920-7. doi: 10.1007/s00535-008-2257-7. Epub 2008 Dec 24. PMID 19107335
- [Background] Pace F, Negrini C, Wiklund I, Rossi C, Savarino V; ITALIAN ONE INVESTIGATORS STUDY GROUP. Quality of life in acute and maintenance treatment of non-erosive and mild erosive gastro-oesophageal reflux disease. Aliment Pharmacol Ther. 2005 Aug 15;22(4):349-56. doi: 10.1111/j.1365-2036.2005.02558.x. PMID 16098002
- [Background] Laine L, DeVault K, Katz P, Mitev S, Lowe J, Hunt B, Spechler S. Vonoprazan Versus Lansoprazole for Healing and Maintenance of Healing of Erosive Esophagitis: A Randomized Trial. Gastroenterology. 2023 Jan;164(1):61-71. doi: 10.1053/j.gastro.2022.09.041. Epub 2022 Oct 10. PMID 36228734
- [Background] Shin JM, Kim N. Pharmacokinetics and pharmacodynamics of the proton pump inhibitors. J Neurogastroenterol Motil. 2013 Jan;19(1):25-35. doi: 10.5056/jnm.2013.19.1.25. Epub 2013 Jan 8. PMID 23350044
- [Background] Abdel-Aziz Y, Metz DC, Howden CW. Review article: potassium-competitive acid blockers for the treatment of acid-related disorders. Aliment Pharmacol Ther. 2021 Apr;53(7):794-809. doi: 10.1111/apt.16295. Epub 2021 Feb 16. PMID 33592125
- [Background] Laine L, Sharma P, Mulford DJ, Hunt B, Leifke E, Smith N, Howden CW. Pharmacodynamics and Pharmacokinetics of the Potassium-Competitive Acid Blocker Vonoprazan and the Proton Pump Inhibitor Lansoprazole in US Subjects. Am J Gastroenterol. 2022 Jul 1;117(7):1158-1161. doi: 10.14309/ajg.0000000000001735. Epub 2022 Mar 16. PMID 35294415
- [Background] Koloski NA, Jones M, Hammer J, von Wulffen M, Shah A, Hoelz H, Kutyla M, Burger D, Martin N, Gurusamy SR, Talley NJ, Holtmann G. The Validity of a New Structured Assessment of Gastrointestinal Symptoms Scale (SAGIS) for Evaluating Symptoms in the Clinical Setting. Dig Dis Sci. 2017 Aug;62(8):1913-1922. doi: 10.1007/s10620-017-4599-6. Epub 2017 May 27. PMID 28551709
- See also: Almutairi MB, Alsulaimi SM, Alghamdi RA, et al. Evaluation of GERD Diagnosis, Management, and Outcomes. The Egyptian Journal of Hospital Medicine. 2018 ;72(9):5195-5202. — https://journals.ekb.eg/article_10741.html